CLINICAL TRIAL: NCT05823402
Title: Use of SPECT-CT for Comparison of Dosimetry Methods in PSMA-targeted Radioligand Therapy (SPECTacular Study)
Acronym: SPECTacular
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BAMF Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BAMF-2022-02
Record Dates: First submitted 2023-04-07; First posted 2023-04-21 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
MeSH Terms: interventions — Single Photon Emission Computed Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SPECT/CT (Experimental): All patients enrolled will undergo 5 additional (6 total) SPECT/CT scans per treatment cycle. Current FDA approved PSMA radioligand therapy is administered over 6 cycles, so there will be a total of 30 additional SPECT/CT scans during this study.
  During each treatment cycle, patients will have a SPECT/CT scan at the following time points after administration of PRLT:
  * 4 Hours
  * 24 Hours (+/- 8 Hours)
  * 48 Hours (+/- 8 Hours)
  * 96 Hours (+/- 8 Hours)
  * 168 Hours (+/- 24 Hours)
  * 336 Hours (+/- 24 Hours)
  Interventions: Diagnostic Test: SPECT/CT

INTERVENTIONS:
Diagnostic Test: SPECT/CT — SPECT/CT imaging can generate 3-dimensional images of the location where the PSMA radioligand therapy has accumulated in the body. SPECT/CT imaging can also measure doses of radiation delivered to those locations.

SUMMARY:
The SPECTacular study will enroll patients who are already undergoing a FDA approved PSMA-targeted Radioligand treatment cycle. During each treatment cycle, patients will receive 5 additional SPECT/CT scans to investigate the limits of agreement between dosimetry (absorbed radiation dose) approximation methods and dosimetry using the triexponential fitting method.

DETAILED DESCRIPTION:
All patients with PSMA-positive tumor and/or Metastases of Prostate Cancer (PSMA-TMPC) who would be undergoing a PSMA-targeted Radioligand Therapy (PRLT) based on independent eligibility criteria for the same, will receive 6 serial SPECT-CT scans for every treatment cycle as a part of our study. The purpose of this investigation is to assess the limits of agreement of commonly employed dosimetry methods used to determine or approximate absorbed doses for organs and tumors compared to a dosimetry method using a triexponential fit requiring 6 post-injection SPECT-CT scans for all treatment cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male, 18 years old or older
4. Histologically or pathologically confirmed prostate adenocarcinoma without predominant small cell component.
5. Patient is receiving PSMA-targeted Radioligand Therapy (PRLT) for treatment of PSMA-positive tumor and/or metastases of prostate cancer. Therapy may be FDA approved or investigational in nature under an approved clinical trial.
6. Ability to lay flat on scanner for duration of SPECT-CT imaging studies (1-2 hours)

Exclusion Criteria:

1. Assessment by the Investigator as unable or unwilling to comply with the requirements of the protocol.
2. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≥ 2
3. All criteria which may preclude a PSMA-radioligand therapy using Lu-177 PSMA-617 or Lu-177 PSMA I&T to be performed as per standardized guidelines and protocols laid down for these treatments and per decision by the treating physician.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Dosimetry Method | Immediately after the completion of SPECT/CT scanning.
  To determine the limits of agreements between dosimetry approximation methods and dosimetry using the triexponential fitting method.

CONTACTS AND LOCATIONS:
Locations (1):
- BAMF Health, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No